CLINICAL TRIAL: NCT05209893
Title: The Effect of Telerehabilitation-Based Exercise and Training Combination on Pain, Function, Balance, Proprioception and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: The Effect of Telerehabilitation-Based Exercise and Training on Outcome Measures in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Serkan Bakırhan, Phd, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24/III
Record Dates: First submitted 2022-01-06; First posted 2022-01-27 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis; Knee Arthritis
Keywords: Gonarthrosis; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (TR) (Experimental): The TR group will be followed up through the application within the 8-week home exercise program.
  Interventions: Other: Telerehabilitation
- Paper Based Rehabilitation (PBR) (Active Comparator): The PBR group will be followed up through the paper instruction within the 8-week home exercise program.
  Interventions: Other: Paper Based Rehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Application based video home exercise for the knee osteoarthritis
  Arms: Telerehabilitation (TR)
Other: Paper Based Rehabilitation — Paper instruction based home exercise for the knee osteoarthritis
  Arms: Paper Based Rehabilitation (PBR)

SUMMARY:
Video exercise component of the telerehabilitation would provide additional contribution to the patients. The aim of this study is to compare the effects of telerehabilitation-based exercise program and conventional (given on paper) exercise and training combination practices on pain, functionality, balance, proprioception and quality of life in patients with knee OA.

DETAILED DESCRIPTION:
Owing to telerehabilitation, exercise video suppliment will enable individuals to learn the exercise programs in the most appropriate way, have comprehensive information about their condition, and communicate easily with their physiotherapists. The aim of this study is to compare the effects of telerehabilitation-based exercise program and conventional (given on paper) exercise and training combination practices on pain, functionality, balance, proprioception and quality of life in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 40 to 65 years
* Being diagnosed with knee osteoarthritis by an orthopedist
* Having a value of 1 or 2 in the Kellgren Lawrence classification
* Having and being able to use the equipment to receive video-based exercise and education support
* Having signed the consent form

Exclusion Criteria:

* Situations that will prevent assessments or communication with the individual
* Knee surgery history
* Having other joint pathologies
* Orthopedic and neurological problems that would prevent evaluation and/or treatment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline Pain at 8 weeks
  On a 10 cm straight line or numerical scale (0: no pain, 10: unbearable pain).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from Baseline Subjective Function at 8 weeks
  WOMAC consists of 3 main headings: pain intensity, stiffness, and physical function. The total score ranges from 0 (no disability) to 96 (complete disability).
Muscle Strength Test with Lafayette Hand Held Dynamometer | Change from Baseline Muscle Strength at 8 weeks
  It is an objective muscle strength measurement tool. Measurements are made 3 times. A rest of 120 seconds is given between measurements. The highest measured value is noted.
Proprioception Measurement with Baseline Bubble Inclinometer | Change from Baseline Proprioception at 8 weeks
  The "absolute angle difference", which is the difference between the targeted angle and the angle realized by the patient in each repetition, is recorded. The arithmetic mean of the absolute angle difference of 3 repetitions is the result data.
Timed Up and Go Test (TUG) | Change from Baseline "Timed Up and Go" test performance at 8 weeks
  Patients are asked to get up from a standard chair, walk 3 meters a safe and comfortable pace, and return without stopping to sit back in the chair safely. The elapsed time is calculated.
Five Times Sit to Stand Test (5TSTS) | Change from Baseline "Five Times Sit to Stand" test performance at 8 weeks
  The test involves patients getting up and sitting again without support from a chair 5 times as soon as possible. Measurements are made with a stopwatch.
3-Meter Backward Walk Test (3MBW) | Change from Baseline "3-Meter Backward Walk" test performance at 8 weeks
  It is determined by measuring a distance of 3 meters. Participants are asked to walk backwards safely but as quickly as possible and stop at the finish line. The time is recorded with a stopwatch.
Modified Four Square Step Test (mFSST) | Change from Baseline "Modified Four Square Step" test performance at 8 weeks
  A suitable ground is divided into four identical squares with a "+" shaped line. Squares are numbered clockwise with numbers 1-4. The patient takes steps on the 1, 2, 3 and 4 squares in sequence without pressing the lines.The test ends when the last foot contact is cut off from the square. The time is recorded with a stopwatch.

SECONDARY OUTCOMES:
EQ-5D-5L | Change from Baseline General Quality of Life at 8 weeks
  The patient is asked to indicate the state of health by marking the most appropriate expression in each of the five dimensions. Index score of the EQ-5D-5L is ranged between 1 to - 0.285. Higher scores indicate better quality of life. VAS score of the EQ-5D-5L is ranged between 0 to 100. Higher scores indicate better quality of life.
Telemedicine Satisfaction Questionnaire | Change from Baseline General Telemedicine Satisfaction at 8 weeks
  This questionnaire consists of 14 items. The level of satisfaction of the patients with the software or system from which they receive treatment or other remote rehabilitation services is evaluated. The tool uses a 5-point Likert scale (1 = strongly disagree, 7 = strongly agree). The total score varies between 14-70 for 14 questions with a maximum of 5 points. Higher scores indicate better satisfaction.
Telehealth Usability Questionnaire | Change from Baseline General Usability Satisfaction at 8 weeks
  The questionnaire consists of 21 items evaluating the distance rehabilitation service. The questionnaire uses a 7-point Likert-type scale (1 = disagree, 7 = agree). The total score is calculated by summing up 21 items.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Principal Investigator — Muğla Sıtkı Koçman University; Cem Yalın Kılınç, MD, Principal Investigator — Muğla Sıtkı Koçman University; Emre Gültaç, MD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tumturk I, Bakirhan S, Ozden F, Gultac E, Kilinc CY. Effect of Telerehabilitation-Based Exercise and Education on Pain, Function, Strength, Proprioception, and Psychosocial Parameters in Patients With Knee Osteoarthritis: A Randomized Controlled Clinical Trial. Am J Phys Med Rehabil. 2024 Mar 1;103(3):222-232. doi: 10.1097/PHM.0000000000002335. Epub 2023 Sep 5. PMID 37678215